CLINICAL TRIAL: NCT02542228
Title: Construction and Validation of a Health-related Quality of Life (HR-QOL) Instrument for Patients With Primary Antibody Deficiency Disease
Brief Title: Construction of a Health-related Quality of Life (HR-QOL) Questionnaire for Patients With Primary Antibody Deficiency Disease
Acronym: HR-QOLPIDD
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: University of Virginia (Other); Boston Children's Hospital (Other); Baylor College of Medicine (Other); Johns Hopkins University (Other); Midwest Immunology Clinic (Unknown); CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: 6119806000
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Immune Deficiency, Antibody
Keywords: Immune Deficiency, antibody; Quality of Life survey
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire survey — The HR-QOL PIDD survey will be administered to the patient by the site PI or the study coordinator. A second survey will be handed to the patient to take home with them and completed at 48-120 hrs. after the clinic visit. The study coordinator will contact the patient during this period to ensure that the patient completes this second survey and returns it to the local study site. A case report form (CRF) of their clinical condition and demographics will be collected at the time of informed consent.

SUMMARY:
This research is being done to construct a survey questionnaire, a quality of life tool, to determine the health, well-being, ability to perform daily activities, and physical, social and emotional functioning in participants with primary immunodeficiency disorders (PIDD). This quality of life (QOL) tool will help physicians understand the effects of PIDD on a person's health. These quality of life surveys are important tools for physicians to measure outcomes for satisfaction and effects of treatment.

DETAILED DESCRIPTION:
A preliminary patient and clinician-generated scale will be validated and modified during a multicenter scale validity study involving 85 patients from 5 sites. Feasibility surveys have been conducted and available sites that can be included in this study include Boston Children's/ Harvard, Midwest Immunology, Johns Hopkins, Children's Hospital at Baylor University, and the University of South Florida at All Children's Hospital Johns Hopkins Medicine. Patients will be enrolled at a clinic non-infusion visit. The purpose of the study will be explained and informed consent obtained. A case report form (CRF) of their clinical condition and demographics will be completed based on the information obtained by the local study coordinator during the interview at the time of the visit. The HR-QOL PIDD survey will be administered to the patient by the site PI or the study coordinator. A second survey will be handed to the patient to take home with them and completed at 48-120 hrs. after the clinic visit. The study coordinator will contact the patient during this period to ensure that the patient completes this second survey and returns it to the local study site. If a patient is on SCIg they will be asked to take the survey 3 days after the SC infusion (if weekly), and complete the paired survey 48-72 hrs later (before another SCIg infusion is scheduled). The study coordinator will obtain an interim history for the period between the paired surveys to ensure that, in general, the condition of the patient has not changed that could invalidate the validation process, and this information will be documented on the addendum case report form (CRF). Patient can return the surveys to the site study coordinator either by mail, fax or electronically by scanning the documents. Paired surveys will be returned to the central study site (USF St Petersburg) for data input.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with documented x-linked agammaglobulinemia, or common variable immunodeficiency, autosomal recessive agammaglobulinemia
2. Subjects must be able to read and speak English
3. Willing to sign consent and follow study schedule.
4. Subjects 18 years to 65 years of age.
5. Subject must be receiving Ig treatment for diagnosis.

Exclusion Criteria:

1. Subject or guardian unwilling to sign consent or adhere to study schedule.
2. Pregnancy,
3. Severe concurrent medical conditions which would prevent treatment or assessment, including significant hematological, renal, lung or liver dysfunction or malignancies
4. Presence of any other medical condition, which in the opinion of the investigator might interfere with performance or interpretation of this study
5. Can not read or understand English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary antibody immune deficiency with x-linked agammaglobulinemia and common variable immune deficiency
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Develop and validate a disease specific Quality of Life Questionnaire for patients with primary antibody immune deficiency disease (PIDD) | one year
  A 28 item questionnaire will be administered to patients with antibody immune deficiency using a 5 point Likert type scale. The questions were generated by clinical immunologist, infusion nurses with feedback from patients. The questions cover all of the SF-36 QOL instrument except body pain. Paired questionnaires were collected 48 to 120 hrs apart from each patient. Rasch analysis will be used to analysis the performance of the questionnaire for disordered items, lack of discrimination between item questions, overlap of questions, and the spread of the 5 point scale that will lead to item reduction. The primary outcome is to generate a validated HR-QOL questionnaire for patients with primary antibody deficiency that will be useful for clinical care and potentially for clinical trials.

REFERENCES:
- [Derived] Ballow M, Conaway MR, Sriaroon P, Rachid RA, Seeborg FO, Duff CM, Bonilla FA, Younger MEM, Shapiro R, Burns TM. Construction and validation of a novel disease-specific quality-of-life instrument for patients with primary antibody deficiency disease (PADQOL-16). J Allergy Clin Immunol. 2017 Jun;139(6):2007-2010.e8. doi: 10.1016/j.jaci.2016.11.029. Epub 2017 Jan 5. No abstract available. PMID 28065678